CLINICAL TRIAL: NCT06481020
Title: Effect of Plant Sterols on Inflammatory, Endothelial Function and Oxidative Stress Markers, Microbiota and Sterol Metabolism in a Cardiovascular Risk Population
Brief Title: Plant Sterols on Cardiovascular Markers, Microbiota and Sterol Metabolism (Cardiofoodsterol)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Hospital Universitario La Fe (Other); University of Bologna (Other)
Responsible Party: Principal Investigator, Guadalupe García Llatas, Principal investigator, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BIONUTEST_2024-0358-1; PID2019-104167RB-I00 (Other Grant/Funding Number: MCIN/AEI/10.13039/501100011033)
Record Dates: First submitted 2024-06-12; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Cardiovascular Diseases; Hypercholesterolemia; Prediabetic State; Overweight and Obesity
Keywords: Cholesterol LDL; Plant Sterols; Inflammation; Oxidative Stress; Microbiota; Sterol Metabolites; Endothelial function; Bioimpedance; Dietary Intake; Physical Activity
MeSH Terms: conditions — Cardiovascular Diseases; Hypercholesterolemia; Prediabetic State; Overweight; Obesity; Inflammation; Motor Activity | interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Supplement (Experimental): PS-containing dietary supplement Sachet containing a powdered microencapsulated free plant sterols (2 g ingredient/day)
  Interventions: Dietary Supplement: Plant sterols 2g/day
- Placebo (Placebo Comparator): Sachet containing the powdered excipients of the dietary supplement
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Plant sterols 2g/day — PS-containing dietary supplement Sachet containing a powdered microencapsulated free plant sterols (2 g ingredient/day) during 8 weeks
  Arms: Dietary Supplement
Dietary Supplement: Placebo — Sachet containing the powdered excipients of the dietary supplement during 8 weeks
  Arms: Placebo

SUMMARY:
Potential cholesterol-lowering effect of a regular intake of a plant sterol (PS)-containing food supplement, in overweight/obese type 1 or 2, normoglycemic/pre-diabetic, with LDL-cholesterol values > 115 mg/dl and not pharmacologically treated participants treated with the PS-containing food supplement or placebo supplement.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death worldwide, with hypercholesterolemia being one of the main risk factors for CVD. The deposition and oxidation of LDL-cholesterol particles triggers a series of molecular events favoring chronic low-grade inflammation, endothelial dysfunction and oxidative stress. This situation promotes atherogenesis thus increasing cardiovascular risk. Obesity favors the secretion of pro-inflammatory mediators and promotes the recruitment of macrophages to adipose tissue, insulin resistance, hyperglycemia and hyperlipidemia, thus increasing the risk of CVD. In addition, obesity has been associated with gut dysbiosis, which in turn is associated with atherosclerosis in some studies. Beneficial effects of PS on LDL-cholesterol and inflammatory, endothelial dysfunction and oxidative stress markers have been reported by several clinical trials. A meta-analysis suggests a lowering effect of PS on body mass index (BMI) in participants with BMI>25. Furthermore, the consumption of PS has been beneficially associated in in vitro studies with changes in intestinal microbial profile, sterol metabolism and short chain fatty acids (SCFA) production. Therefore, the hypothesis is if the consumption of PS as a food supplementation could reduce cardiovascular risk. The present study aims to evaluate the LDL-cholesterol serum levels after regular intake of a food supplement containing PS (2 g/day) in overweight/obese type 1 or 2 patients, normoglycemic /pre-diabetic and with LDL-cholesterol values > 115 mg/dl not pharmacologically treated. This is a crossover study with 21 participants (intake of a food supplement containing PS) and 21 participants (intake of excipient-based placebo), with a first intervention period of 8 weeks. After a 6-week washout period, the treatments are switched, with a second intervention period of 8 weeks. In addition, to the LDL-cholesterol lowering assessment, other biochemical, hematological, inflammatory, endothelial dysfunction and oxidative stress parameters are assessed in serum samples. Moreover, sterol and metabolite profiling in serum and feces, microbiota modulation, anthropometric measurements and body composition, bioimpedance, dietary intake and physical activity questionnaire are evaluated. All parameters are evaluated at the beginning (weeks 0 and 14) and at the end of each intervention period (weeks 8 and 22).

ELIGIBILITY:
Inclusion Criteria:

* BMI: 27-29.9 or 30-39.9
* Plasmatic glucose: < 100mg/dl or 100-125mg/dl
* Glycosylated hemoglobin: < 5.7 or 5.7-6.4
* LDL cholesterol > 115mg/dL
* Serum levels of biochemical and hematological parameters and fat-soluble vitamins within reference ranges.

Exclusion Criteria:

* Subjects on cholesterol-lowering pharmacological treatment
* Smokers
* Alcohol consumption above 30 g/day
* Pregnant or lactating women
* Any infection, serious illness or co-morbidity that may affect the bioavailability of PS (e.g., malabsorption, celiac disease, allergies or food intolerances)
* Diseases of the gastrointestinal tract
* Antibiotic, hormonal or anabolic treatment
* Participants consuming foods enriched with PS or food supplements that contain PS
* Participants who follow specialist weight loss diets, vegans or vegetarians

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Changes in plasmatic LDL-c | 0, 8, 14 and 22 weeks
  LDL-c, calculated by the Friedewald's formula, with repeated measures (at the beginning and at the end of each period the intervention)

SECONDARY OUTCOMES:
Changes in plasmatic total cholesterol | 0, 8, 14 and 22 weeks
  Total cholesterol, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of each period the intervention)
Changes in plasmatic HDL-c | 0, 8, 14 and 22 weeks
  HDL-c, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of each period the intervention)
Changes in plasmatic non-HDL cholesterol | 0, 8, 14 and 22 weeks
  Non-HDL cholesterol, calculated by subtracting HDL-c from total cholesterol, with repeated measures (at the beginning and at the end of each period the intervention)
Changes in plasmatic triglycerides | 0, 8, 14 and 22 weeks
  Triglycerides, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of each period the intervention)
Changes in plasmatic Apo A | 0, 8, 14 and 22 weeks
  Apo A, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of each period the intervention)
Changes in plasmatic Apo B | 0, 8, 14 and 22 weeks
  Apo B, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of each period the intervention
Changes in plasmatic fibrinogen | 0, 8, 14 and 22 weeks
  Fibrinogen, assessed by Clauss coagulometric method, with repeated measures (at the beginning and at the end of each period the intervention)
Changes in plasmatic High-sensitivity C-reactive protein (hsCRP) | 0, 8, 14 and 22 weeks
  hs CRP, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of each period the intervention)
Changes in plasmatic glucose | 0, 8, 14 and 22 weeks
  Glucose, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of each period the intervention)
Changes in plasmatic insulin | 0, 8, 14 and 22 weeks
  Insulin, assessed by enzymatic-colorimetric methods, with repeated measures (at the beginning and at the end of each period the intervention
Changes in plasmatic Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | 0, 8, 14 and 22 weeks
  HOMA-IR, calculated by mathematical formula from the fasting insulin and fasting glucose levels, with repeated measures (at the beginning and at the end of each period the intervention)
Changes in serum levels of the sterols and metabolites profile | 0, 8, 14 and 22 weeks
  Profile sterols and metabolites, assessed by gas chromatography coupled with flame ionization detector (GC-FID), with repeated measures (at the beginning and at the end of each period the intervention)
Changes in feces levels of the sterols and metabolites profile | 0, 8, 14 and 22 weeks
  Profile sterols and metabolites, assessed by gas chromatography coupled with flame ionization detector (GC-FID), with repeated measures (at the beginning and the end of each period the intervention)
Changes in serum interleukin 10 (IL-10) | 0, 8, 14 and 22 weeks
  IL-10, assessed by immunochemical techniques, with repeated measures (at the beginning and the end of each period the intervention)
Changes in serum interleukin 12p70 (IL-12p70) | 0, 8, 14 and 22 weeks
  IL-12p70, assessed by immunochemical techniques, with repeated measures (at the beginning and the end of each period the intervention)
Changes in serum interleukin 1β (IL-1β) | 0, 8, 14 and 22 weeks
  IL-1β, assessed by immunochemical techniques, with repeated measures (at the beginning and the end of each period the intervention)
Changes in serum interleukin 6 (IL-6) | 0, 8, 14 and 22 weeks
  IL-6, assessed by immunochemical techniques, with repeated measures (at the beginning and the end of each period the intervention)
Changes in serum interleukin 8 (IL-8) | 0, 8, 14 and 22 weeks
  IL-8, assessed by immunochemical techniques, with repeated measures (at the beginning and the end of each period the intervention)
Changes in serum tumor necrosis factor alpha (TNFα) | 0, 8, 14 and 22 weeks
  TNFα, assessed by immunochemical techniques, with repeated measures (at the beginning and the end of each period the intervention)
Changes in serum vascular cell adhesion molecule-1 (VCAM-1) | 0, 8, 14 and 22 weeks
  VCAM-1, assessed by immunochemical techniques, with repeated measures (at the beginning and the end of each period the intervention)
Changes in serum E-Selectin | 0, 8, 14 and 22 weeks
  E- Selectin, assessed by immunochemical techniques, with repeated measures (at the beginning and the end of each period the intervention)
Changes in serum endothelin (ET-1) | 0, 8, 14 and 22 weeks
  ET-1, assessed by immunochemical techniques, with repeated measures (at the beginning and the end of each period the intervention
Changes in serum plasminogen activator inhibitor-1(PAI-1) | 0, 8, 14 and 22 weeks
  PAI-1, assessed by immunochemical techniques, with repeated measures (at the beginning and the end of each period the intervention)
Changes in plasmatic LDL-cholesterol oxidation | 0, 8, 14 and 22 weeks
  LDL-cholesterol oxidation, assessed by enzyme kits, with repeated measures (at the beginning and the end of each period the intervention)
Changes in plasmatic 8-isoprostane | 0, 8, 14 and 22 weeks
  8-isoprostane, assessed by enzyme kits, with repeated measures (at the beginning and the end of each period the intervention)
Changes in plasmatic malondialdehyde (MDA) | 0, 8, 14 and 22 weeks
  MDA, assessed by ultra-performance liquid chromatography-MS (UPLC-MS), with repeated measures (at the beginning and the end of each period the intervention
Changes in reduced glutathiones (GSH) | 0, 8, 14 and 22 weeks
  GSH, assessed by ultra-performance liquid chromatography-MS (UPLC-MS), with repeated measures (at the beginning and the end of each period the intervention)
Changes in oxidized glutathione (GSSG) | 0, 8, 14 and 22 weeks
  GSSG, assessed by ultra-performance liquid chromatography-MS (UPLC-MS), with repeated measures (at the beginning and the end of each period the intervention)
Changes in the composition of microbiota in feces | 0, 8, 14 and 22 weeks
  Composition of microbiota, assessed by genetic sequencing and subsequent biostatistical analysis, with repeated measures (at the beginning and the end of each period the intervention)
Changes in feces of short-chain fatty acids (SCFAs) | 0, 8, 14 and 22 weeks
  SCFAs, assessed by high-performance liquid chromatography with an ultraviolet detector (HPCL-UV), with repeated measures (at the beginning and the end of each period the intervention)
Changes in plasmatic levels of cholesterol oxidation products (COPs) | 0, 8, 14 and 22 weeks
  COPs, assessed by gas chromatography-mass spectrometry, with repeated measures (at the beginning and the end of each period the intervention)
Changes in body weight (WT) | 0, 8, 14 and 22 weeks
  WT, assessed by standard balance scale, with repeated measures (at the beginning and the end of each period the intervention)
Changes in body height (HT) | 0, 8, 14 and 22 weeks
  HT, assessed by tape measure, with repeated measures (at the beginning and the end of each period the intervention)
Changes in body circumferences | 0, 8, 14 and 22 weeks
  Circumferences, assessed by tape measure, with repeated measures (at the beginning and the end of each period the intervention)
Changes in Bioelectrical impedance analysis (BIA) | 0, 8, 14 and 22 weeks
  BIA, assessed by bio-impedance meter, with repeated measures (at the beginning and the end of each period the intervention)
Assessment of dietary intake | 0, 8, 14 and 22 weeks
  Food frequency survey Questionnaire (FFQ) is used, consisting in 136 questions divided into the different food groups (dairy products; eggs, meat and fish; vegetables; fruit; pulses and cereals; oils and fats; bakery and confectionery; miscellaneous; drinks) indicating the average frequency of consumption during the past year, which can be scored as never or almost never, per month (1-3), per week (1, 2-4,5-6), per day (1, 2-3, 4-6, 6+), with repeated of questionnaire (at the beginning and the end of each period the intervention)
Evaluation of the physical activity to measure quality of life | 0, 8, 14 and 22 weeks
  International physical activity questionnaire-short form (IPAC-SF) is used, consisting in 7 questions. Intensity, frequency and duration of the exercise are evaluated through metabolic equivalent of task (METs). This allows to differentiate 3 levels of physical activity:
  Low: Not enough activity to achieve the next level
  Moderate: 3 or more days of vigorous physical activity for at least 20 minutes per day, 5 or more days of moderate physical activity and/or walking at least 30 minutes per day, or 5 or more days of any combination of walking, moderate or vigorous physical activity achieving at least a total of 600 METs.
  High: Vigorous physical activity at least 3 days per week achieving a total of a least 1500 METs, or 7 days of any combination of walking, with moderate and/or vigorous physical activity, achieving a total of a least 3000 METs.
  With repeated of questionnaire (at the beginning and the end of each period the intervention)
Evaluation of the Mediterranean diet adherence to measure quality of life | 0, 8, 14 and 22 weeks
  Mediterranean diet adherence screener (MEDAS) is used, consisting in 14 questions (each one 0 or 1 point, final score between 0 and 14). Results are ranged between 0-7 points (low adherence), 7-10 (moderate adherence), and 10-14 (high adherence) With repeated of questionnaire (at the beginning and the end of each period the intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe Garcia Llatas, Professor, Principal Investigator — University of Valencia
Locations (1):
- Hospital Universitario y Politécnico La Fe de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanco-Morales V, Garcia-Llatas G, Yebra MJ, Sentandreu V, Lagarda MJ, Alegria A. Impact of a Plant Sterol- and Galactooligosaccharide-Enriched Beverage on Colonic Metabolism and Gut Microbiota Composition Using an In Vitro Dynamic Model. J Agric Food Chem. 2020 Feb 19;68(7):1884-1895. doi: 10.1021/acs.jafc.9b04796. Epub 2019 Sep 26. PMID 31523960
- [Background] Blanco-Morales V, Silvestre RLA, Hernandez-Alvarez E, Donoso-Navarro E, Alegria A, Garcia-Llatas G. Influence of Galactooligosaccharides on the Positive Effect of Plant Sterol-Enriched Beverages on Cardiovascular Risk and Sterol Colon Metabolism. J Agric Food Chem. 2022 Jan 19;70(2):532-542. doi: 10.1021/acs.jafc.1c06120. Epub 2022 Jan 11. PMID 35012310
- [Background] Caudet J, Trelis M, Cifre S, Tapia G, Soriano JM, Rodrigo R, Merino-Torres JF. Do Intestinal Unicellular Parasites Have a Role in the Inflammatory and Redox Status among the Severely Obese? Antioxidants (Basel). 2022 Oct 23;11(11):2090. doi: 10.3390/antiox11112090. PMID 36358463
- [Background] Heggen E, Kirkhus B, Pedersen JI, Tonstad S. Effects of margarine enriched with plant sterol esters from rapeseed and tall oils on markers of endothelial function, inflammation and hemostasis. Scand J Clin Lab Invest. 2015 Apr;75(2):189-92. doi: 10.3109/00365513.2014.992040. Epub 2015 Jan 1. PMID 25553599
- [Background] Oliveira Godoy Ilha A, Sutti Nunes V, Silva Afonso M, Regina Nakandakare E, da Silva Ferreira G, de Paula Assis Bombo R, Rodrigues Giorgi R, Marcondes Machado R, Carlos Rocha Quintao E, Lottenberg AM. Phytosterols Supplementation Reduces Endothelin-1 Plasma Concentration in Moderately Hypercholesterolemic Individuals Independently of Their Cholesterol-Lowering Properties. Nutrients. 2020 May 22;12(5):1507. doi: 10.3390/nu12051507. PMID 32455866
- [Background] Mannarino E, Pirro M, Cortese C, Lupattelli G, Siepi D, Mezzetti A, Bertolini S, Parillo M, Fellin R, Pujia A, Averna M, Nicolle C, Notarbartolo A. Effects of a phytosterol-enriched dairy product on lipids, sterols and 8-isoprostane in hypercholesterolemic patients: a multicenter Italian study. Nutr Metab Cardiovasc Dis. 2009 Feb;19(2):84-90. doi: 10.1016/j.numecd.2008.03.012. Epub 2008 Aug 31. PMID 18762410
- [Background] Menendez-Carreno M, Steenbergen H, Janssen HG. Development and validation of a comprehensive two-dimensional gas chromatography-mass spectrometry method for the analysis of phytosterol oxidation products in human plasma. Anal Bioanal Chem. 2012 Feb;402(6):2023-32. doi: 10.1007/s00216-011-5432-2. Epub 2011 Oct 5. PMID 21972006